CLINICAL TRIAL: NCT06599125
Title: Risk Factors of Mortality in Neonatal Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hossam El-deen Kheder, 71515, Assuit, Assiut University
Other Study IDs: neonatal pneumonia
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neonatal pneumonia, a lower chest infectious disease, is one of the most serious and fatal diseases in young infants.(1) Neonates may catch pneumonia vertically from mother or horizontally from the environment at birth time.

DETAILED DESCRIPTION:
Neonatal pneumonia, a lower chest infectious disease, is one of the most serious and fatal diseases in young infants. Neonates may catch pneumonia vertically from mother or horizontally from the environment at birth time. Time of catching infection can be classified into:

Prenatal; that's intrauterine, it is also called Congenital Pneumonia. The pathogen may investigate the neonatal lung intrauterine through chrioamniotic membranes or trans-placental.

At birth, during the first week after birth Early onset pneumonia, however pathogen mat be from intrauterine or at birth canal; and mostly this type of pneumonia is bacterial.

After the first week of life late onset pneumonia. It is common to be of nosocomial or community acquired.

Neonatal Pneumonia is the second leading cause of death after neonatal sepsis. It accounts for 152,000 to 490,000 of infants aged < 1 year annually, Research papers reported that in 2016, 2.6 million neonatal deaths were reported representing a global burden of 19 neonatal deaths per 1000 live births and in 2017 the annual neonatal mortality rate NMR was highest in east, west and central Africa. About specific-cause-mortality of these estimations, lower chest infection represented 13.5% of these deaths, and had the highest incidece in the first 28 days of life in live birth.

In the majority of cases, causing pathogen of neonatal pneumonia is viral, however community and hospital acquired pneumonia are frequently bacterial that caused by Haemophilus influenzae, Streptococcus agalactiae or Enterobacteriaceae species. Although pneumonia occurs in all ages, neonatal pneumonia is associated with comorbidities and mortality in age below 59 days.

Lung of newborn is volurnable to pneumonia due to variable risk factors. Some of these factors are attributed to mother, other to neonate and the rest is to labor circumstances. In general, neonate is suseptabile to infection due to weak immunity; a factor that is more potentiating in premature neonate. However, maternal risk factors resulting in congenital pneumonia are for example represented in systemic diseases, infection during pregnancy as toxoplasmosis, cytomegalovirus CMV, herpes simplex virus HSV. Neonates catch early onset pneumonia in perinatal duration whether before labor through placenta, ascending infection intrauterine or from pathogens in birth canal during vaginal delivery. Late onset pneumonia is due to exposure to the pathogen in community, although, a common risk factor for late onset pneumonia is low birth weight and prematurity.Reported factors that potentiate mortality in case pneumonia are living in developing countries, drining infested water, maternal smoking, late starting of treatment and the more younger of child the higher risk they are in.

Diagnosis of neonatal pneumonia is difficult in neonates because they may experience no symptoms, or have symptoms that are part of other syndromes unlike older children or adults that have clear symptoms. In this study we aim to evaluate the clinical, laboratory, radiological and other risk factors that predict mortality in term and preterm 32 to 36 weeks neonates admitted with pneumonia in neonatalogy unit in Assuit university Children hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn aged ≤ 30 days (0 to 30d.)
2. Neonates diagnosed with pneumonia during the first month of life.

Exclusion Criteria:

1. Infant aged more than one month.
2. Neonates with ches x-ray negative for pneumonia.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Risk factors of mortality in neonatal pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Methods | Baseline
  Our study will be retrospective cross sectional study,and the cases will be collected from archive of neonatology unit of assiut university children hospital as well as prospective single group cohort study and will be conducted in neonatalogy unit in Children Hospital in Assiut University for one year duration. Newborn babies aged since birth to ≤ 28 days who have been diagnosed with pneumonia will be included.
History | Baseline
  Full history will be taken from all patient with emphasis on the following :
  Maternal history:
  Demographic history
  1- Maternal age
  3-- socioeconomic state
  Medical conditions:
  Any infection during pregnancy. Events during pregnancy (e.g. PROM, pre-eclampsia, Gestationale diabetes, …). Autoimmune diseases. Any comorbid disease that affect immunity (DM, CKD, etc. …).
  Surgical history:
  Any operation conducted during pregnancy. Blood transfusion (during pregnancy).
  Obstetric history:
  Mode of labor ( Cesarean / Vaginal). Maternal fever Parity.
  Neonatal history:
  Time of diagnosis (prenatal- at birth- first day- second day- … - 30th day) Signs of hypoxia at birth (cyanosis- respiratory distress- ……) Tachypnea Fever Admission in NICU
Examination | Baseline
  General and local examination will be done to all patient with emphasis on the following:
  Oxygen saturation. Temperature. Centeral and Peripheral Cyanosis. Congenital anomalies.
  Chest examination:
  Inspection:
  Deformity of thorax. / Shape of the thorax (Deformity, Movement,…) Signs of distress (tachypnea, nasal flaring, Lower chest indrawing). Respiratory rate Palpation Percution
  Auscultation:
  Breathing sounds. Decreased air entry Rales or ronchi Crepitation
Investigations | Baseline
  All patients will be subjectd to the following investigations:
  Complete blood count (CBC) for neonate. Chest X-ray. Blood culture. C- reactive protein. ESR Serum Na, K. Kidney Function Test (KFT) Liver Function Test (LFT)
  Some of cases will be subjectd to the following investigations according to the clinical status :
  CT - Chest Echocardiograpgy Bronchoalveolar lavage Neonatal Pneumonia Mortality will be considered as death occurring in pneumonic neonate during their first month of life while hospitalization.
Sample size | Baseline
  Based on determining the main outcome variable, The estimated minimum required sample size is 85 patients .
  The sample size was calculated using Epi-info version 7 software, based on the following assumptions:Main outcome variable is aim to evaluate the clinical, laboratory, radiological and other risk factors that predict mortality in term and preterm (32 to 36 weeks) neonates admitted with pneumonia in neonatalogy unit in Assuit university Children hospital.Based on previous studies (7), The prevalence of neonatal pneumonia in Egypt varies by region and study. In a study conducted at Qena University Hospital, neonatal pneumonia was found in 17.2% of neonates admitted with respiratory diseases and based on the percentage confidence limits of 5% and a Confidence level=80% .

REFERENCES:
- [Background] North K, Frade Garcia A, Crouch M, Kimsen S, Hoey A, Wade C, Kim Y, Chou R, Edmond KM, Lee ACC, Rees CA. Efficacy of Antibiotic Regimens for Pneumonia in Young Infants Aged 0-59 Days: A Systematic Review. Pediatrics. 2024 Aug 1;154(Suppl 1):e2024066588G. doi: 10.1542/peds.2024-066588G. PMID 39087803
- [Background] Hug L, Alexander M, You D, Alkema L; UN Inter-agency Group for Child Mortality Estimation. National, regional, and global levels and trends in neonatal mortality between 1990 and 2017, with scenario-based projections to 2030: a systematic analysis. Lancet Glob Health. 2019 Jun;7(6):e710-e720. doi: 10.1016/S2214-109X(19)30163-9. PMID 31097275
- [Result] Baseer KAA, Mohamed M, Abd-Elmawgood EA. Risk Factors of Respiratory Diseases Among Neonates in Neonatal Intensive Care Unit of Qena University Hospital, Egypt. Ann Glob Health. 2020 Feb 26;86(1):22. doi: 10.5334/aogh.2739. PMID 32140431